CLINICAL TRIAL: NCT05510336
Title: Assessment of Concentric Needle Technique for the Management of Temporomandibular Joint Internal Derangement Randomized Controlled Trial (RCT)
Brief Title: Assessment of Concentric Needle Technique in Temporomandibular Joint (TMJ) Internal Derangement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Hassan Mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Concentric needle technique
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: TMJ Disc Disorder
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Concentric needle technique TMJ arthrocentesis using lactated ringer solution to help reduce inflammatory mediators and anterior disc discplacement with reduction
  Interventions: Procedure: Arthrocentesis
- Control group (Active Comparator): Double needle technique TMJ arthrocentesis using lactated ringer solution to help reduce inflammatory mediators and anterior disc discplacement with reduction
  Interventions: Procedure: Arthrocentesis

INTERVENTIONS:
Procedure: Arthrocentesis — Injection of lactated ringer solution in the TMJ to wash out inflammatory mediators and help reducing anterior disc displacement with reduction

SUMMARY:
The aim of the study is to evaluate the effectivenes of using two concentric needles in comaprsion with the normal traditional two distant needles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age ranges from 18-60.
2. Patients with painful clicking.
3. Patients free of systemic conditions that might affect the TMJ or interfere with carrying out the surgical procedure (osteoarthritis, rheumatoid arthritis, uncontrolled diabetes).

Exclusion Criteria:

1. Patients out of the specified range group
2. Patients with painless TMJ clicking.
3. Patients with osteo-arthritic changes of the TMJ.
4. Patients with systemic conditions that might affect the TMJ or interfere with carrying out the surgical procedure (osteoarthritis, rheumatoid arthritis, uncontrolled diabetes).
5. Patients with previous TMJ surgeries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain felt during the procedure TMJ arthrocentesis | baseline
  Visual analogue scale from zero to ten (zero indicates no pain and ten indicates worst pain)

DOCUMENTS (1):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05510336/Prot_000.pdf